CLINICAL TRIAL: NCT05798130
Title: Assessment of Oxygen Extraction Rate Changes Following Red Blood Cell Transfusion in the Intensive Care Unit: a Prospective Observational Non-interventional Study
Brief Title: Assessment of Oxygen Extraction Rate Changes Following Red Blood Cell Transfusion in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ahmet Salih Tüzen, MD, Medical Doctor, Izmir Katip Celebi University
Other Study IDs: 2023-GOKAE-0103
Record Dates: First submitted 2023-03-03; First posted 2023-04-04 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-11

CONDITIONS: Red Blood Cell Transfusion; Oxygen Consumption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oxygen Extraction Rate < 30% Group: Oxygen Extraction Rate < 30%
  Interventions: Other: No intervention group.
- Oxygen Extraction Rate ≥ 30% Group: Oxygen Extraction Rate ≥ 30%
  Interventions: Other: No intervention group.

INTERVENTIONS:
Other: No intervention group. — No intervention group.

SUMMARY:
Restrictive and liberal approaches to hemoglobin targets are used when deciding on red blood cell transfusions in patients who do not have acute bleeding and have a hemodynamically stable course in the intensive care unit. However, physiologic trigger points that assess tissue oxygenation when deciding on blood transfusion in patients are also among the important topics of study in recent years. In this study, the investigators will evaluate the oxygen extraction rate, which is an important indicator of the balance between tissue oxygen delivery and consumption. Whether oxygen extraction rate can be used as a trigger for blood transfusion will be determined by clinical outcomes in ICU patients. If physiologic transfusion targets are feasible, the risks of unnecessary transfusions can be avoided with individualized targets, and the decision to transfuse blood can be made without delay in patients requiring red blood cell transfusion.

DETAILED DESCRIPTION:
This study will be prospective and observational in the Intensive Care Unit of Izmir Katip Celebi University Atatürk Training and Research Hospital. The study will not include any intervention and intervention groups. The study will enroll patients who have no acute bleeding, are hemodynamically stable, have been followed in the ICU for at least 24 hours, have a central venous catheter, and for whom the decision to transfuse red blood cells has been made according to the critical care protocol. Informed consent is obtained from the patient or first-degree relatives.

No additional procedures will be performed on patients during the study, and the decision to transfuse will not be influenced by the results of the examinations. For patients in whom the decision to transfuse red blood cells was made in accordance with the critical care protocol, the clinical decision and policy to transfuse a single unit and, accordingly, a restrictive transfusion strategy with a target hemoglobin of 7 g/dl are applied.

The patient's oxygen extraction rate is calculated using the following formula by considering the difference between the oxygen content of the venous and arterial blood gasses measured before transfusion.

CaO2 = SaO2 x Hb x 1.39 + (PaO2 x 0.0031) CcvO2 = ScvO2 x Hb x 1.39 + (PcvO2 x 0.0031) O2ER = CaO2 - CcvO2/CaO2

Patients to be followed until day 90 post-transfusion will be evaluated in two separate groups according to oxygen extraction rate < 30% and ≥30% after pretransfusion blood gas analysis. The primary objective of the study is to evaluate the percentage change in oxygen extraction rate after transfusion between the two groups with oxygen extraction rates of < 30% and ≥30%. The secondary objective is to examine the difference between the groups in 28-day mortality, near-infrared spectroscopy (NIRS) values related to tissue oxygenation, amount of blood products consumed, and length of ICU stay, as well as complication rates such as acute renal failure and acute lung injury.

Age, sex, comorbidities, reasons for ICU hospitalization, and number of days in the ICU before transfusion of participants are demographically recorded. The following values will be noted by the observer before and after transfusion: systolic blood pressure, mean arterial pressure, heart rate, NIRS values, blood gas analysis; pH, PaO2, PaCO2, SaO2, base deficit, HCO3, lactate, PcvO2, PcvCO2, ScvO2, FiO2, CaO2, CcvO2, AV-O2 difference, O2ER, PaO2/FiO2, lactate clearance, CVP, vasoactive inotrope score. In addition, the SAPS, APACHE-II, SOFA scores of the 1st and 5th day, hemoglobin and hematocrit values of the first 5 days, MCV, MPV, RDW, INR, platelet count, blood urea nitrogen, creatinine, number of mechanical ventilator-dependent days, number of vasopressor-dependent days, and number of the intensive care unit stay days are monitored. In addition, the development of complications such as acute respiratory failure, acute renal failure, development of infections, stroke, and myocardial infarction in participants will be tracked. The occurrence of mortality at day 7, 28, and 90 will be reported in the study results.

In the reference study1, patients were studied in 2 separate groups with oxygen extraction rates of < 30% and ≥30%. There was a significant difference between the groups in terms of change in oxygen extraction rate after 15 minutes. The mean±standard deviation of the groups was -5.2±7.8 and 0.7±5.8, respectively, and p=0.004. In the power analysis performed, it was assumed that the type 1 error was 0.05 and the power of the study was 0.80, so it would be sufficient to reach 29 patients in both groups. Considering a 10% probability of loss to data acquisition, it would be sufficient to reach a total of 65 patients.

All statistical analyzes will be performed using the SPSS 22 program. Descriptive statistics are expressed with mean and standard deviation for continuous variables and with numbers and percentages for categorical variables. Prior to all analyzes, skewness- kurtosis tests, normality tests, and histogram graphs are used to determine whether the data conform to the normal distribution. In determining differences in means between groups, the T test for independent variables or the T test for dependent variables is used for variables with normal distribution; the Mann-Whitney U test or the Wilcoxon test is used for variables that do not conform to normal distribution. The chi-square test or the Fischer exact test is used to determine the differences between groups for categorical variables. The difference values between the means of repeated measures in the groups are evaluated using the Mann-Whitney U test. In the case of more than two time periods, the evaluation of time, groups, and joint effects is performed with the two-way test ANOVA (analysis of variance) for repeated measures. Post-hoc analyzes will be performed using the Bonferonni test. The effect of independent variables on mortality is assessed by logistic regression analysis. Kaplan-Meier survival curves will be analyzed with respect to the oxygen extraction rate predicting 28-day mortality in both groups. For all analyzes to be performed, a p< 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients followed in the intensive care unit for at least 24 hours
* Patients with central venous catheters
* Patients who have received a decision to transfuse red blood cells

Exclusion Criteria:

* Patients with hemodynamically unstable
* Patients with acute bleeding
* Patients in hemorrhagic shock
* Patients with acute traumatic brain injury
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage change in oxygen extraction rate | After transfusion of 15.minutes
  Evaluate the percentage change in oxygen extraction rate after and before red blood cell transfusion between the two groups with oxygen extraction rates of > 30% and ≥30%.

SECONDARY OUTCOMES:
7, 28 and 90 days mortality | 7, 28 and 90 days
  7, 28 and 90 days mortality
Near infrared spectroscopy values change | After transfusion of 15.minutes
  Near infrared spectroscopy values change
Length of ICU stay | up to 90 days
  Length of ICU stay
Complication rates | up to 90 days
  Complication rates
Length of hospital stay | up to 90 days
  Length of hospital stay
Number of mechanical ventilation dependent days | up to 90 days
  Number of mechanical ventilation dependent days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Salih Tüzen, Principal Investigator — Izmir Katip Celebi University Ataturk Training and Research Hospital, Department of Anesthesiology and Reanimation; Murat Aksun, Principal Investigator — Izmir Katip Celebi University Ataturk Training and Research Hospital, Department of Anesthesiology and Reanimation
Locations (1):
- Izmir Katip Celebi University Ataturk Training and Research Hospital, Department of Anesthesiology and Reanimation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Orlov D, O'Farrell R, McCluskey SA, Carroll J, Poonawala H, Hozhabri S, Karkouti K. The clinical utility of an index of global oxygenation for guiding red blood cell transfusion in cardiac surgery. Transfusion. 2009 Apr;49(4):682-8. doi: 10.1111/j.1537-2995.2008.02022.x. PMID 19347976
- [Derived] Tuzen AS, Aksun M, Sencan A, Girgin S, Golboyu BE, Kirbas G, Sanli O. Assessment of oxygen extraction rate changes following red blood cell transfusion in the intensive care unit: A prospective observational noninterventional study. Transfusion. 2025 May;65(5):863-875. doi: 10.1111/trf.18164. Epub 2025 Mar 25. PMID 40134137
- [Derived] Tuzen AS, Aksun M, Sencan A, Girgin S, Golboyu BE, Kirbas G, Sanli O. Assessment of oxygen extraction rate changes following red blood cell transfusion in the intensive care unit: a protocol for a prospective observational non-interventional study. BMJ Open. 2023 Aug 30;13(8):e074413. doi: 10.1136/bmjopen-2023-074413. PMID 37648379